CLINICAL TRIAL: NCT03785912
Title: Randomized Controlled Trial (RCT) to Evaluate the Efficacy and Cost-effectiveness of an Internet-based Self-help Program for People With Adjustment Problems After an Accident
Brief Title: SelFIT: Internet-based Treatment for Adjustment Problems After an Accident
Acronym: SelFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss Accident Insurance Fund SUVA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01059
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Adjustment Impairment; Accident; Adjustment Disorders; Mental Disorder
MeSH Terms: conditions — Adjustment Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based self-help (Experimental): The self-help program consists of eight text- and video-based modules. All participants in this group receive immediate access to the self-help program. The program's self-management approach does not provide for regular support from a specialist. However, participants can contact the study team if they need or want additional help.
  Interventions: Behavioral: Internet-based self-help
- Waiting control group (No Intervention): Access to internet-based intervention after 12 weeks.

INTERVENTIONS:
Behavioral: Internet-based self-help — Eight cognitive-behavioral, mindfulness and acceptance commitment based modules focusing on different aspects of adjustment problems after having an accident.
  Arms: Internet-based self-help

SUMMARY:
In this study, people who suffer from adjustment problems after having experienced an accident will be randomized to one of two study groups. The first group receives access to the internet-based self-help intervention immediately. The second group is a waiting control group that receives access to the program 12 weeks later. In both conditions additional care or treatment is allowed. The aim of the study is to investigate the efficacy and cost-effectiveness of an internet-based self-help intervention for people with adjustment problems after an accident compared to a waiting list. There are 6 assessments, which all take place online: baseline, two between-measurements (after 4 and 8 weeks), post assessment (after 12 weeks) and two follow-up assessments (after 3 and 6 months). All participants from both groups are asked to fill out all assessments.

ELIGIBILITY:
Inclusion Criteria: All participants must...

* be at least 18 years old
* give a declaration of consent to participate in the study
* have access to the Internet
* understand and master the German language to the degree that they understand the contents and instructions of the study
* exceed the cut-off value for at least a mild psychological burden on the depression-anxiety stress scale (DASS- 21)
* be able to specify an emergency address in the event of an acute crisis
* have experienced and can specify an accident during a period of two weeks to two years prior to participation in the current study that lead to the conditions described above.

Exclusion Criteria: Excluded are persons who...

* show severe depressive symptoms (Beck depression inventory [BDI-II] > 29)
* show suicidal tendencies (BDI-II Suicide item > 1)
* have a known diagnosis of psychotic or bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
DASS-21: Depression, Angst, Stress-Skala (Lovibond & Lovibond, 1995) | 7 minutes
  21-item questionnaire assessing depression, anxiety and stress symptoms

SECONDARY OUTCOMES:
BDI-II:Beck Depression Inventory (Beck et al., 1996; Margraf & Ehlers, 1998) | 5-10 minutes
  21-item questionnaire assessing depressive symptoms
ADNM-20: Adjustment Disorder - New Module 20 (Lorenz et al., 2016) | 6 minutes
  20-item questionnaire assessing adjustment disorder symptoms and severity
SF-12: Short Form Health Survey (Ware et al., 1996) | 5 minutes
  12-item questionnaire assessing various aspects of well-being
LOT-R: Revised Life Orientation Test (Herzberg et al., 2006) | 3 minutes
  10-item questionnaire assessing optimism and pessimism
BVI: Berner Verbitterungsinventar (Znoj, 2008) | 3 minutes
  18-item questionnaire assessing embitterment
FAB: Fragebogen Arbeit und Wohlbefinden (Abegglen et al., 2017) | 5 minutes
  24-item questionnaire assessing different aspects of work- and health-related topics
TIC-P: Treatment inventory of Costs in Psychiatric Patients (Bouwmans et al., 2013) | 20 minutes
  58-item questionnaire assessing costs related to an accident
ZUF-8: Zufriedenheitsfragebogen (Attkisson & Zwick, 1982) | 2 minutes
  8-item questionnaire assessing content with an online-program
SUS: System Usability Scale (Brooke, 1996) | 3 minutes
  10-item questionnaire assessing usability of an online-program
SWE: Skala zur Allgemeinen Selbstwirksamkeit (Jerusalem & Schwarzer, 2003) | 3 minutes
  10-item questionnaire assessing general self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Hansjörg Znoj, Prof. Dr., Study Director — University of Bern; Thomas Berger, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- Universität Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hegy JK, Brog NA, Berger T, Znoj H. Web-based Self-help Program for Adjustment Problems After an Accident (SelFIT): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 17;9(12):e21200. doi: 10.2196/21200. PMID 33331830